CLINICAL TRIAL: NCT03657719
Title: Open-labeled(Part 1), Single-group(Part 2), Randomized(Part 2), Double-blind(Part 2), Active-controlled(Part 2) Pharse II Clinical Trial to Evaluate Safety and Efficacy(Immunogenicity) of GC3114 in Elderly Healthy Subjects
Brief Title: A Study to Evaluate the Safety and Efficacy(Immunogenicity) of GC3114 in Elderly Healthy Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GC3114_P2
Record Dates: First submitted 2018-08-27; First posted 2018-09-05 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Part 1 : Single group, Part2 : Parallel group
Who Masked: Participant, Investigator
Masking Description: Part 1 : Open label, Part 2 : Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GC3114 (Experimental): Pre-filled syringe inj., 0.5ml, Once, IM
  Interventions: Biological: GC3114
- Active Comparator: GCFLU Quadrivalent (Active Comparator): Pre-filled syringe inj., 0.5ml, Once, IM
  Interventions: Biological: GCFLU Quadrivalent

INTERVENTIONS:
Biological: GC3114 — High-dose Quadrivalent influenza vaccine
  Arms: GC3114
Biological: GCFLU Quadrivalent — Quadrivalent influenza vaccine
  Arms: Active Comparator: GCFLU Quadrivalent

SUMMARY:
Elderly healthy subjects will be once administered GC3114A(High-dose Quadrivalent influenza vaccine) or GCFLU Quadrivalent Pre-filled syringe inj..

DETAILED DESCRIPTION:
Elderly healthy subjects will be once administered GC3114A(High-dose Quadrivalent influenza vaccine) or GCFLU Quadrivalent Pre-filled syringe inj..

Safety and immunological efficacy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged over 65 years old
* Informed consent form has been signed and dated

Exclusion Criteria:

* Known systemic hypersensitive to eggs, chicken proteins, or any of the vaccine components
* Personal history of Guillain-Barre syndrome(GBS)
* Subjects with severe chronic disease who are considered by investigator to be ineligible for the study
* Subjects who received a vaccination within 28 days before enrollment or who are scheduled for another vaccination during the study
* Immunocompromised subjects with immunodeficiency disease or subjects receiving immunosuppressive or immunomodulating therapy

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
Adverse Event | for 7 days from Day0/during study period
  Solicited/Unsolicited Adverse Event

SECONDARY OUTCOMES:
Percentage of participants achieving pre-defined Seroconversion Before and following vaccination | Day 0 and Day 28
  Seroconversion rate (SCR)
Percentage of participants achieving pre-defined Seroprotection Before and following vaccination | Day 0 and Day 28
  Seroprotection rate (SPR)
Geometric Mean Titer of Antibodies to the Investigational Product Before and Following vaccination | Day 0 and Day 28
  Geometric Mean Titer(GMT)
Geometric Mean Ratio of Antibodies to the Investigational Product Before and Following vaccination | Day 0 and Day 28
  Geometric Mean Ratio(GMR)

CONTACTS AND LOCATIONS:
Overall Officials: Woo Joo KIm, M.D, Ph.D, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea